CLINICAL TRIAL: NCT00028171
Title: Pharmacokinetics of Tacrolimus in Kidney Transplant Recipients: Once Daily Versus Twice Daily Dosing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0824
Record Dates: First submitted 2001-12-17; First posted 2001-12-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus

SUMMARY:
Tacrolimus is a medication given to transplant patients to help prevent rejection. The purpose of this study is to see if tacrolimus can be taken once a day instead of twice a day in kidney transplant patients.

Transplant patients are required to take several medications to prevent rejection and to treat complications after their transplantation. Because of the complicated dosing schedule, it can be difficult for patients to follow their medication schedule. Taking fewer medications less frequently may help transplant patients to better manage their drug therapy.

Tacrolimus is better absorbed in the body if it is taken in the morning than if it is taken in the evening. This suggests that tacrolimus can be taken once every morning instead of twice daily in order to produce appropriate drug exposure to prevent organ rejection without increased side effects.

ELIGIBILITY:
Inclusion Criteria: 1) Kidney transplant recipients (18 years or older) at Washington University/Barnes Hospital taking tacrolimus-based immunosuppression; 2) Stable kidney transplant recipients (>6 months post-transplantation, serum creatinine < 2 ml/dL, no history of rejection); 3) Stable immunosuppression (therapeutic tacrolimus concentrations, no change in tacrolimus dose within one month prior to the study); 4) Subjects must agree to abstain from alcohol and caffeine for 48 hours prior to the pharmacokinetics studies.

Exclusion Criteria: 1) Pregnant women or nursing mothers; 2) Patients unwilling or unable to comply with the protocol; 3) Significant liver impairment (AST or ALT > 2 x upper limit of normal, or total bilirubin > upper limit of normal); 4) Anemia: Hematocrit < 30%; 5) Use of concomitant P450 3A4/p-glycoprotein inducers or inhibitors; 6) Current smoking; 7) Patients with diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University/Barnes Jewish Hospital, St Louis, Missouri, United States